CLINICAL TRIAL: NCT06168786
Title: A Phase II, Single-arm, Open-label, Multi-Centers Study of Cadonilimab Combined With Fruquintinib and SBRT as A Third-line and Posterior Line Treatment in Patients With MSS Colorectal Cancer
Brief Title: Cadonilimab Combined With Fruquintinib and SBRT as Athird-line and Posterior Line Treatment in Patients With MSS CRC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xianglin Yuan, Huazhong University of Science and Technology, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRC-II-001
Record Dates: First submitted 2023-12-05; First posted 2023-12-13 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — HMPL-013

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cadonilimab plus Fruquintinib and SBRT (Experimental)
  Interventions: Drug: Fruquintinib; Drug: Cadonilimab; Radiation: SBRT

INTERVENTIONS:
Drug: Fruquintinib — Fruquintinib:5mg ,qd,po, d1-d14, q3w
Drug: Cadonilimab — Cadonilimab:10mg/kg, ivgtt, d1, q3w
Radiation: SBRT — SBRT:8-10Gy×5F，qod， in 10 days

SUMMARY:
A Phase II Study to Assess the Efficacy and Safety of Cadonilimab Combined With Fruquintinib and SBRT as A third-line and Posterior Line Treatment in Patients With MSS Colorectal Cancer

ELIGIBILITY:
Inclusion Criteria:

* Provision of written Informed Consent Form (ICF) prior to any study specific procedures
* Age ≥ 18 years, ≤75 years
* Histologically or cytologically confirmed advanced Stage IV primary colorectal cancer
* MSI status: MSS
* At least two or more standard systemic therapies prior treatment (based on Fu, oxaliplatin, irinotecan, bevacizumab and cetuximab) of cytotoxic chemotherapy, treatment failure or intolerable toxicities
* ECOG 0-1
* Patients must have measurable lesions
* Expected overall survival ≥12 weeks
* AST, ALT and alkaline phosphatase ≤ 2.5 times the upper limit of normal (ULN)，Serum bilirubin ≤ 1.5 x ULN，creatinine<ULN
* Prothrombin time (PT), international standard ratio (INR) ≤1.5 × ULN
* Patients are allowed to have received radiotherapy, but the time from entering the group must be more than 4 weeks, and the currently selected radiotherapy lesions and evaluable lesions must be lesions that have not received radiotherapy
* Fertile male or female patients voluntarily used an effective contraceptive method during the study period and within 6 months of the last study medication

Exclusion Criteria:

* Patients have received anti-PD-1 / PD-L1 or anti-CTLA-4 immunotherapy or other immunoexperimental drugs
* Patients with severe autoimmune diseases: active inflammatory bowel disease (including Crohn's disease and ulcerative colitis), rheumatoid arthritis, scleroderma, systemic lupus erythematosus, autoimmune vasculitis (such as Wegener's granuloma), etc
* Symptomatic interstitial lung disease or active infection/non-infectious pneumonia
* Risk factors of intestinal perforation: active diverticulitis, abdominal abscess, gastrointestinal obstruction, abdominal cancer or other known risk factors of intestinal perforation
* If the patients underwent surgery, they should wait for the wound to heal completely before being considered for enrollment
* History of other malignant tumors（(except for the cured localized tumors, such as skin basal cell carcinoma, skin squamous cell carcinoma, superficial bladder carcinoma, prostate carcinoma in situ, cervical carcinoma in situ, and breast carcinoma in situ）
* Patients who are preparing for or have previously received an organ or allogeneic bone marrow transplant
* Moderate or severe ascites with clinical symptoms required therapeutic puncture, drainage or Child-Pugh score >2 (except those who only show a small amount of ascites on imaging without clinical symptoms); Uncontrolled or moderate or higher pleural effusion or pericardial effusion
* History of gastrointestinal bleeding or a definite tendency to gastrointestinal bleeding within 6 months before the start of treatment
* Abdominal fistula, gastrointestinal perforation, or abdominal abscess developed within 6 months before the start of study treatment
* Known hereditary or acquired bleeding (e.g. coagulation dysfunction) or thrombotic tendencies, e.g. in hemophiliacs; Currently or recently (within 10 days prior to the start of study therapy) used full dose oral or injectable anticoagulants or thrombolytic agents for therapeutic purposes (allowing prophylactic use of low-dose aspirin, low molecular weight heparin)
* Aspirin (> 325 mg / day (maximum antiplatelet dose) or dipyridamole, ticlopidine, clopidogrel (≥ 75 mg) and cilostazol are currently used or have been used recently (within 10 days before the start of study treatment)
* Thrombosis or embolism events such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction) and pulmonary embolism occurred within 6 months before the start of the study
* Patient with an active infection, heart failure, heart attack, unstable angina pectoris, or unstable arrhythmia within the last 6 months
* Physical examination or clinical trial findings that the investigator believes may interfere with the results or put the patient at increased risk for treatment complications, or other uncontrollable diseases
* The researchers believe that the patient has a lesion and needs emergency palliative radiotherapy / emergency surgery (spinal cord compression, brain hernia, pathological fracture)
* Lactating or pregnant women
* History of immunodeficiency, including HIV positive, other acquired or congenital immunodeficiency diseases, or organ transplantation
* Patients with mental illness, substance abuse, or social problems that affect compliance will not be enrolled after researcher's review
* Known active infection and active tuberculosis infection were not included in the group; However, patients with hepatitis B virus (HBV) and hepatitis C virus (HCV) infection can be included in the group if their condition is stable after antiviral treatment
* Patients who received live vaccine within 30 days prior to enrollment
* Have clinical symptoms or diseases of the heart that are not well controlled
* Systolic blood pressure > 140mmHg or diastolic blood pressure > 90mmHg regardless of any antihypertensive drugs； or a history of hypertensive crisis or hypertensive encephalopathy
* Major vascular disease (such as aortic aneurysms requiring surgical repair or recent peripheral arterial thrombosis) developed within 6 months
* Severe, unhealed or open wounds and active ulcers or untreated fractures
* Received major surgery within 4 weeks prior to the start of study treatment (except for diagnosis) or expected to require major surgery during the study period
* Inability to swallow tablets, malabsorption syndrome or any condition affecting gastrointestinal absorption
* Had a history of intestinal obstruction and/or had clinical signs or symptoms of gastrointestinal obstruction within 6 months prior to initiation of study therapy, including incomplete obstruction related to pre-existing disease or requiring routine parenteral hydration, parenteral nutrition, or tube feeding
* Patients with signs/symptoms of incomplete obstruction/obstructive syndrome/ileus at initial diagnosis may be admitted to the study if they have received definitive (surgical) treatment to resolve symptoms
* There is evidence of abdominal gas accumulation that cannot be explained by puncture or recent surgical procedures
* Metastatic disease involving a major airway or blood vessel or a large mediastinal tumor mass located in the center (<30 mm from the crest)
* Patients with a history of hepatic encephalopathy
* For those who currently have interstitial pneumonia or interstitial lung disease, or who have a history of interstitial pneumonia or interstitial lung disease requiring hormone therapy, Or other subjects with pulmonary fibrosis, institutionalized pneumonia, pneumoconiosis, drug-related pneumonia, idiopathic pneumonia that may interfere with the judgment and management of immune-related pulmonary toxicity, or with evidence of active pneumonia or severe impairment of lung function visible on chest CT during the screening period, radiation pneumonia is allowed in the radiation field; Active tuberculosis
* Presence of active autoimmune disease or history of autoimmune disease with possible recurrence; Participants with non-systemic skin diseases such as vitiligo, psoriasis, and alopecia, controlled type 1 diabetes treated with insulin, or asthma in complete remission in childhood, were enrolled without any intervention as adults; Patients with asthma who require medical intervention with bronchodilators are not included
* Use of immunosuppressants or systemic hormone therapy for immunosuppression within 14 days prior to initiation of study therapy
* Known history of severe allergy to any monoclonal antibody, anti-angiogenesis targeting drug
* Severe infection, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia, in the 4 weeks prior to initiation of study treatment; Therapeutic antibiotics were given orally or intravenously within 2 weeks prior to the start of study therapy
* According to the investigator's judgment, the patient has other factors that may affect the study results or lead to the forced termination of the study. There are serious abnormalities in laboratory examination, accompanied by family or social factors, which will affect the safety of the patient

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-06-20 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | up to 42 months
  To assess the efficacy of Cadonilimab Combined With Fruquintinib and SBRT for patients with advanced colorectal cancer by assessment of progression free survival (PFS) using Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1).

SECONDARY OUTCOMES:
Objective response rate (ORR) | up to 42 months
  CR + PR rate according to the RECIST version 1.1 guidelines.
Disease control rate (DCR) | up to 42 months
  Disease control rate (DCR):CR + PR + SD rate according to the RECIST version 1.1 guidelines.
Overall survival (OS) | until death
  The time interval between the start date of study drug and the date of death (any cause)
quality of life (QOL) | up to 42 months
  QOL according to QOL-C30
AEs | up to 42 months
  Adverse reactions refer to the occurrence and development of diseases in the process of using drugs according to normal usage and dosage to prevent, diagnose or treat diseases.Adverse reactions unrelated to the purpose of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No